CLINICAL TRIAL: NCT01439815
Title: A Single-Center, Randomized, Double-Masked, Placebo-Controlled Evaluation of the Efficacy of Flonase (Fluticasone Propionate Nasal Spray) Compared to Placebo Nasal Spray in the Allergen BioCube (ABC) Model
Brief Title: An Allergen BioCube (ABC) Study Evaluating the Efficacy of Fluticasone Propionate Nasal Spray Compared to Placebo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 11-100-0007
Record Dates: First submitted 2011-09-19; First posted 2011-09-23 (Estimated); Results first posted 2021-03-24 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2020-11

CONDITIONS: Allergic Rhinitis; Allergic Conjunctivitis
MeSH Terms: conditions — Rhinitis, Allergic; Conjunctivitis, Allergic | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Nasal Spray (Placebo Comparator): Two sprays in each nostril daily starting the day in office on Day 0 for up to a 17 day period until Day 16.
  Interventions: Drug: Saline Nasal Spray
- Fluticasone Propionate (Active Comparator): Two sprays in each nostril daily starting the day in office on Day 0 for up to a 17 day period until Day 16.
  Interventions: Drug: Fluticasone Propionate Nasal Spray

INTERVENTIONS:
Drug: Fluticasone Propionate Nasal Spray — two sprays in each nostril once daily
  Other Names: Flonase
  Arms: Fluticasone Propionate
Drug: Saline Nasal Spray — two sprays in each nostril once daily
  Arms: Placebo Nasal Spray

SUMMARY:
The purpose of this study is to evaluate the onset of action of fluticasone propionate nasal spray compared to placebo nasal spray in reducing nasal allergic signs and symptoms following ragweed exposure in the Allergen BioCube (ABC) after up to 14 days of at home dosing.

ELIGIBILITY:
Inclusion Criteria:

* provide written informed consent and signed HIPAA form;
* be able and willing to follow all instructions and attend the study visits;
* if female and of childbearing potential, be not pregnant, nursing or planning a pregnancy, be willing to submit a pregnancy test at Visit 1 and at exit visit, and to use adequate method of birth control
* have a positive history of seasonal allergic rhinitis to ragweed;
* have a positive skin test reaction to ragweed of within the past 24 months;
* manifest sufficient allergic rhinitis symptoms during ragweed exposure in the ABC

Exclusion Criteria:

* known intolerance or allergy to antihistamines or corticosteroids;
* have a compromised lung function at Visit 1;
* develop a compromised lung function at Visits 2-6
* have any presence of active sinus or nasal infection at any visit;
* have experienced an acute upper or lower respiratory tract infection or acute sinusitis within 30 days of visit 1;
* have significant nasal anatomical deformities or any condition that does not allow subject to breathe through the nose (includes, but is not limited to: septal deviation, septal perforations, nasal polyps, rhinitis medicamentosa)
* have had any nasal surgical intervention in the past;
* have a known history of glaucoma
* have planned surgery (nasal, ocular or systemic) during the trial period or within 30 days thereafter;
* inability or refusal to discontinue contact lens wear during all visits;
* use disallowed medications during the study or appropriate pre-study washout period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Shazly, MD, Principal Investigator — ORA, Inc.
Locations (1):
- Ora, Inc., Andover, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from one site in the US.
Pre-assignment Details: Twenty-two participants enrolled and completed the study. Participant flow and baseline characteristics are presented for the 22 subjects that met all inclusion criteria, none of the exclusion criteria and were randomized to receive Fluticasone Propionate or Placebo nasal spray twice daily based on the randomization list.
Groups:
- Fluticasone Propionate Nasal Spray; Placebo Nasal Spray: Two sprays in each nostril daily starting the day in office on Day 0 for up to a 17 day period until Day 16.
Period: Overall Study
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Started | 11 | 11
All Randomized Participant Population | 11 | 11
Completed | 11 | 9
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Nasal Signs and Symptoms Score From Baseline (Day 0) to Visit 5 (Day 16)
Description: The change in the total sum of the four symptoms (total nasal symptom scores - TNSS) ranging from 0 to 16 with higher score indicating a more severe reaction.
  The change in the TNSS score between Day 0 and Day 16 was analyzed.
Time Frame: pre-ABC exposure and approximately every 15 minutes, up to 180 minutes, while in the ABC on Day 0 and Day 16
Population: All Randomized Participants Population - All participants who received study treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 11 | 11
units on a scale
  pre-ABC | -0.7 (1.8) | 0.3 (1.8)
  15 minutes | -2.8 (3.4) | 0.9 (3.8)
  30 minutes | -4.1 (3.4) | -0.6 (3.0)
  45 minutes | -3.9 (4.2) | -0.3 (3.1)
  60 minutes | -4.7 (3.6) | -0.9 (3.3)
  75 minutes | -4.5 (4.5) | -2.3 (3.7)
  90 minutes | -4.5 (4.3) | -1.7 (3.3)
  105 minutes | -5.0 (4.0) | -1.6 (2.5)
  120 minutes | -5.9 (3.1) | -0.7 (3.5)
  135 minutes | -4.8 (4.0) | -0.5 (3.2)
  150 minutes | -5.3 (3.6) | -1.7 (2.6)
  165 minutes | -5.4 (3.2) | -1.6 (2.8)
  180 minutes | -5.9 (3.0) | -0.6 (3.0)

2. Secondary Outcome: Change in Baseline Nasal Itching Score on Day 0 to Average Nasal Itching Score on Day 16
Description: Nasal Itching was assessed by the participants pre-ABC exposure and approximately every 15 minutes while in the ABC on Day 0 and Day 16 on a 0-4 scale (0 = none to 4 = severe). The change in average nasal itching score between Day 0 and Day 16 was analyzed.
Time Frame: pre-ABC exposure and approximately every 15 minutes, up to 180 minutes, while in the ABC on Day 0 and Day 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 11 | 11
units on a scale
  Pre-ABC | -0.2 (0.6) | 0.1 (0.7)
  15 minutes | -1 (1) | 0.3 (0.8)
  30 minutes | -1 (1.2) | -0.1 (0.6)
  45 minutes | -0.8 (1.6) | -0.1 (0.9)
  60 minutes | -1.3 (1.3) | -0.3 (0.9)
  75 minutes | -1.3 (1.5) | -0.5 (0.8)
  90 minutes | -1 (1.6) | -0.6 (0.7)
  105 minutes | -1.3 (1.3) | -0.5 (0.8)
  120 minutes | -1.5 (1.1) | -0.4 (0.8)
  135 minutes | -1.5 (1.2) | -0.3 (0.8)
  150 minutes | -1.5 (1.3) | -0.2 (0.8)
  165 minutes | -1.5 (1.1) | -0.2 (1)
  180 minutes | -1.8 (1.2) | 0 (1.1)

3. Secondary Outcome: Change in Baseline Sneezing Score on Day 0 to Average Sneezing Score on Day 16
Description: Sneezing was assessed by the participants pre-ABC exposure and approximately every 15 minutes while in the ABC on Day 0 and Day 16 on a 0-4 scale (0 = none to 4 = severe). The change in average sneezing score between Day 0 and Day 16 was analyzed.
Time Frame: pre-ABC exposure and approximately every 15 minutes, up to 180 minutes, while in the ABC on Day 0 and Day 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 11 | 11
units on a scale
  Pre-ABC | -0.1 (0.3) | 0.2 (0.9)
  15 minutes | -0.5 (1.1) | 0.1 (0.9)
  30 minutes | -0.9 (0.8) | -0.4 (0.8)
  45 minutes | -0.9 (1.1) | 0 (0.9)
  60 minutes | -1.3 (1.1) | -0.2 (1)
  75 minutes | -1.1 (1.3) | -0.6 (1.3)
  90 minutes | -1.1 (1.4) | -0.3 (1.2)
  105 minutes | -1.2 (1.1) | -0.4 (1)
  120 minutes | -1.3 (1.3) | -0.1 (1.1)
  135 minutes | -0.9 (1.4) | 0 (0.9)
  150 minutes | -0.8 (1.3) | -0.7 (1)
  165 minutes | -1.1 (0.9) | -0.6 (1)
  180 minutes | -1.2 (0.8) | -0.1 (0.7)

4. Secondary Outcome: Change in Baseline Rhinorrhea Score on Day 0 to Average Rhinorrhea Score on Day 16
Description: Rhinorrhea was assessed by the participants pre-ABC exposure and approximately every 15 minutes while in the ABC on Day 0 and Day 16 on a 0-4 scale (0 = none to 4 = severe). The change in average rhinorrhea score between Day 0 and Day 16 was analyzed.
Time Frame: pre-ABC exposure and approximately every 15 minutes, up to 180 minutes, while in the ABC on Day 0 and Day 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 11 | 11
units on a scale
  Pre-ABC | -0.4 (0.8) | 0 (0.5)
  15 minutes | -0.9 (0.9) | 0.4 (1.2)
  30 minutes | -1.5 (0.8) | 0 (0.8)
  45 minutes | -1.1 (1.1) | -0.2 (1)
  60 minutes | -1.2 (1) | -0.1 (1)
  75 minutes | -1.3 (1.1) | -0.7 (1.3)
  90 minutes | -1.5 (1) | -0.5 (1.1)
  105 minutes | -1.4 (1.4) | -0.5 (1)
  120 minutes | -1.7 (0.6) | -0.1 (1)
  135 minutes | -1.4 (1.1) | 0 (1.1)
  150 minutes | -1.5 (0.8) | -0.4 (0.8)
  165 minutes | -1.4 (0.8) | -0.4 (0.8)
  180 minutes | -1.5 (0.9) | -0.3 (1.2)

5. Secondary Outcome: Change in Baseline Nasal Congestion Score on Day 0 to Average Nasal Congestion Score on Day 16
Description: Nasal Congestion was assessed by the participants pre-ABC exposure and approximately every 15 minutes while in the ABC on Day 0 and Day 16 on a 0-4 scale (0 = none to 4 = severe). The change in average nasal congestion score between Day 0 and Day 16 was analyzed.
Time Frame: pre-ABC exposure and approximately every 15 minutes, up to 180 minutes, while in the ABC on Day 0 and Day 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 11 | 11
units on a scale
  Pre-ABC | -0.1 (1) | 0 (0.7)
  15 minutes | -0.4 (1.2) | 0.1 (1.3)
  30 minutes | -0.7 (1.3) | -0.1 (1.2)
  45 minutes | -1.1 (1.1) | 0 (0.9)
  60 minutes | -1 (1.1) | -0.4 (0.8)
  75 minutes | -0.9 (1.1) | -0.5 (1)
  90 minutes | -1.1 (1.2) | -0.3 (0.9)
  105 minutes | -1.2 (1) | -0.2 (0.9)
  120 minutes | -1.5 (0.9) | -0.2 (0.9)
  135 minutes | -1.1 (1.1) | -0.2 (0.9)
  150 minutes | -1.4 (0.9) | -0.3 (0.8)
  165 minutes | -1.4 (0.9) | -0.3 (0.8)
  180 minutes | -1.5 (0.9) | -0.1 (0.9)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline (Day 0) through study completion (Day 16). All subjects who received study medication were evaluable for the safety analysis.
Description: Throughout the visits, staff collected all Adverse Events reported, elicited, or observed.
Groups:
- Fluticasone Propionate Nasal Spray; Placebo Nasal Spray: Two sprays in each nostril daily starting the day after Day 1 for up to 14 days.
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 1/11 | 3/11
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluticasone Propionate Nasal Spray (N=11) | Placebo Nasal Spray (N=11)
hives (neck) (General disorders) | 0 (0) | 1 (1)
dizziness (General disorders) | 1 (1) | 0 (0)
headache (General disorders) | 0 (0) | 1 (1)
hives (face) (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes